CLINICAL TRIAL: NCT03871543
Title: Late Night Study 2: End-of-Day Assessment of Asymptomatic and Symptomatic Soft Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR-6290
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Part 1 (Other): All eligible subjects enrolled into Part 1 will be fit and dispensed with Test Lens 1
  Interventions: Device: AquaComfort Plus
- Part 2 (Other): All eligible subjects (based on CLDEQ responses) enrolled into Part 2 will be fit and dispensed with Test Lens 2 and will follow the same procedures as Part 1.
  Interventions: Device: Acuvue Oasys 1-Day

INTERVENTIONS:
Device: AquaComfort Plus — Test Lens 1
  Arms: Part 1
Device: Acuvue Oasys 1-Day — Test Lens 2
  Arms: Part 2

SUMMARY:
This is a 2-Part, 8-Visit, single-center, open-label, bilateral and dispensing clinical study. In Part 1 (Visits 1-4) all subjects will be Test Lens 1, in Part 2 (Visits 1-4) eligible subjects will be dispensed Test Lens 2 based on their responses to the CLDEQ-8 questionnaire. Subjects scoring between 11 and 19 on the CLDEQ will not continue into Part 2

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the criteria listed to be enrolled in the study.

  1. They are 18-45 years of age (inclusive).
  2. They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
  3. They are willing and able to follow the protocol.
  4. They agree not to participate in other clinical research while enrolled on this study.
  5. They currently use daily disposable soft daily wear contact lenses (worn bilaterally) (within the last six months) which may be spherical, toric or multifocal.
  6. They agree to wear their lenses for at least 12-14 hours per day.
  7. They own a wearable pair of spectacles (by self-report).
  8. They have a spherical contact lens prescription in the range +6.00 to -10.00 DS (based on the calculated ocular refraction).
  9. They have up to a maximum of 1.00 DC of refractive astigmatism (based on the calculated ocular refraction).
  10. They have best corrected distance visual acuity of at least 0.20 binocularly

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. They have an ocular disorder which would normally contraindicate contact lens wear.
  2. They have a systemic disorder which would normally contraindicate contact lens wear.
  3. No ocular topical medications (including comfort drops) from 24 hours prior to study visits or during the wear of any study lenses.
  4. They are regularly using anti-inflammatory or pain medications (i.e. medication routinely used more than twice per week).
  5. They have had cataract surgery.
  6. They have had corneal refractive surgery.
  7. They are pregnant or breast-feeding.
  8. They have any infectious disease (e.g. hepatitis) or any immunosuppressive disease (e.g. HIV) or a history of anaphylaxis or severe allergic reactions.
  9. They are an employee or immediate family member of an employee of the clinical site (e.g. Investigator, Coordinator, Technician).
  10. They have taken part in any other clinical trial or research within two weeks prior to starting this study.
  11. History of allergy to sodium fluorescein or lissamine green.
  12. They have any corneal distortion e.g. as a result of previous rigid lens wear or have keratoconus.
  13. They any slit lamp findings of Efron Grade 3 or greater (e.g. corneal edema, corneal neovascularization, tarsal abnormalities, conjunctival injection) or findings of < Grade 3 which in the investigator's opinion would contraindicate contact lens wear.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (1):
- The University of Manchester - Eurolens Research, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 196 subjects were enrolled into this study. Of those enrolled, 184 subjects were dispensed at least one study lens while, 12 subjects failed to meet all eligibility criteria. Of those dispensed, 46 completed the study and 138 subjects were discontinued.
Groups:
- Test 1 (Dailies Aqua Comfort Plus) \ Test 2 (Acuvue Oasys 1-Day): All eligible subjects in this study were first the dispensed Test 1 (Dailies Aqua Comfort Plus) lens during the first period and the Test 2 (Acuvue Oasys 1-Day) lens during the second period
Period: Period 1
Arm/Group | Test 1 (Dailies Aqua Comfort Plus) \ Test 2 (Acuvue Oasys 1-Day)
Started | 184
Completed | 48
Not Completed | 136
Not completed — Unsatisfactory Lens Fitting due Test Article | 10
Not completed — Investigator Error | 1
Not completed — Protocol Violation | 2
Not completed — COVID-19 Related | 1
Not completed — Subject No Longer meets Eligibility Criteria | 112
Not completed — Withdrawal by Subject | 10
Period: Period 2
Arm/Group | Test 1 (Dailies Aqua Comfort Plus) \ Test 2 (Acuvue Oasys 1-Day)
Started | 48
Completed | 46
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed at least one study lens.
Groups:
- Asymptomatic: Subjects with a Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) score less than or equal to 10 after 2-week wears of lens wear.
- Symptomatic: Subjects with a Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) score greater than or equal to 20 after 2-week wears of lens wear.
- Other: Subjects with a Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) score between 11-19 after 2-week wears of lens wear.
- Unknown: Subjects with Unknown Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) score
- Total: Total of all reporting groups
Arm/Group | Asymptomatic | Symptomatic | Other | Unknown | Total
Number analyzed (Participants) | 88 | 20 | 58 | 18 | 184
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28 (6.67) | 27.8 (7.09) | 25.1 (6.32) | 28.1 (8.83) | 27.1 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 16 | 45 | 11 | 134
  Male | 26 | 4 | 13 | 7 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 9 | 5 | 23 | 8 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 4 | 0 | 13
  White | 69 | 13 | 27 | 10 | 119
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 4 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Lid Margin Staining (Part1: Dailies Aqua Comfort Plus)
Description: Lid margin staining of the upper and lower eyelids was performed in the left eye (OS) only using lissamine green. The following attributes were graded subjectively for each eyelid: Horizontal length of staining (Grade 0: < 2mm, Grade 1: 2-4 mm, Grade 2: 5-9 mm, Grade 3: >9 mm), and Sagittal width of staining relative to width of wiper (Grade 0: <25%, Grade 1: 25-50 %, Grade 2: 51-75%, Grade 3: >75%). The Average staining grade for each eyelid was also calculated which is the average of the horizontal and sagittal grades. Higher Lid Margin Staining values indicate that more staining was observed.
Time Frame: 14 Hours Follow-up at Visit 4
Population: All subjects who successfully complete all visits and do not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 28 | 18
Number analyzed (Eyes) | 28 | 18
Units on a Scale
  Upper Lid | 1.02 (0.822) | 1.25 (0.943)
  Lower Lid | 1.45 (0.896) | 1.78 (0.988)
Statistical Analysis 1: Comparison: Asymptomatic vs Symptomatic; Upper Lid; Test type: Other — Statistical Difference; Mixed Models Analysis; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean difference = 0.159, 95% CI 1-sided [lower limit -0.402], Standard Error of Mean 0.287 — Mean difference was calculated as Symptomatic minus Asymptomatic
Statistical Analysis 2: Comparison: Asymptomatic vs Symptomatic; Lower Lid; Test type: Other — Statistical Difference; Mixed Models Analysis; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean Difference = 0.236, 95% CI 1-sided [lower limit -0.328], Standard Error of Mean 0.289 — Mean difference was calculated as Symptomatic minus Asymptomatic

2. Primary Outcome: Non-invasive Tear Break-up Time (Part1: Dailies Aqua Comfort Plus)
Description: NIBUT was measured in timed seconds using the Medmont topographer for the right eye (OD) only. NIBUT values are positive, where higher NIBUT times (seconds) indicate a more stable tear film.
Time Frame: 14 Hours Follow-up at Visit 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Seconds
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 28 | 18
Number analyzed (Eyes) | 28 | 18
Seconds | 4.43 (3.386) | 4.32 (3.613)
Statistical Analysis 1: Comparison: Asymptomatic vs Symptomatic; Test type: Other — Statistical difference; Generalized Linear Mixed Model; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean Ratio = 0.918, 95% CI 1-sided [upper limit 1.227] — Mean ratio was calculated as Symptomatic divided by Asymptomatic

3. Primary Outcome: Tear Meniscus Height (Part1: Dailies Aqua Comfort Plus)
Description: The lower tear meniscus in the right eye (OD) only was imaged and measured in mm using optical coherence tomography (OCT). Lower TMH values indicate reduced tear quantity.
Time Frame: 14 Hours Follow-up at Visit-4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 28 | 18
Number analyzed (Eyes) | 28 | 18
mm | 0.20 (0.058) | 0.19 (0.069)
Statistical Analysis 1: Comparison: Asymptomatic vs Symptomatic; Test type: Other — Statistical difference; Mixed Models Analysis; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean Difference = -0.010, 95% CI 1-sided [upper limit 0.022], Standard Error of Mean 0.019 — Mean difference was calculated as Symptomatic minus Asymptomatic

4. Primary Outcome: Tear Film Osmolarity (Part1: Dailies Aqua Comfort Plus)
Description: Tear film osmolarity were collected and measured in (mOsms/L) in the right eye (OD) only using the Tearlab (Tearlab Corp.).Higher tear osmolarity values may be associated with ocular dryness. Participants were classified as symptomatic or asymptomatic based on their subjective questionnaire responses for the CLDEQ-8 questionnaire assessed after two weeks of lens wear (Visit 2). CLDEQ-8 is a validated patient-reported outcome measure assessing patient-experience of symptoms relating to contact lens dryness.
Time Frame: 14 Hours Follow-up at Visit 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mOsms/L
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 28 | 18
Number analyzed (Eyes) | 28 | 18
mOsms/L | 299.00 (12.098) | 301.89 (12.107)
Statistical Analysis 1: Comparison: Asymptomatic vs Symptomatic; Test type: Other — Statistical difference; Mixed Models Analysis; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean Difference = 1.185, 95% CI 1-sided [lower limit -4.613], Standard Error of Mean 3.483 — Mean difference was calculated as Symptomatic minus Asymptomatic

5. Primary Outcome: Number of White Blood Cells Per Frame in Eyelid Margin (Part1: Dailies Aqua Comfort Plus)
Description: Images, using Confocal Microscopy were taken in both eyes for both the upper and lower eyelid in the central lid area. These images were used to determine the mean density of inflammatory white blood cells. Higher white blood cell counts may be associated with an increased inflammatory response. The number of white blood cells is a count of the number of cells 'per frame'. A frame has a fixed area of 400 x 400 microns. The average number of White Blood Cells was reported for each group.
Time Frame: 2-Week Follow-up (after 6 hours lens wear) at Visit 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of white blood cells per frame
Units Other Than Participants: Eyes
Arm/Group | Asymptomatic | Symptomatic
Number analyzed (Participants) | 28 | 18
Number analyzed (Eyes) | 56 | 34
number of white blood cells per frame
  Upper Lid | 7.94 (8.450) | 14.91 (12.562)
  Lower | 5.89 (6.184) | 12.19 (12.210)
Statistical Analysis 1: Comparison: Asymptomatic vs Symptomatic; Upper Lid; Test type: Other — Statistical difference; Generalized Linear Mixed Model; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean Ratio = 1.984, 95% CI 1-sided [lower limit 1.198] — Mean Ratio was calculated as Symptomatic divided by Asymptomatic
Statistical Analysis 2: Comparison: Asymptomatic vs Symptomatic; Lower Lid; Test type: Other — Statistical Difference; Generalized Linear Mixed Model; The Kenward and Roger Method was used for the denominator degrees of freedom; Mean Ratio = 1.800, 95% CI 1-sided [lower limit 1.093] — Mean Ratio was calculated as Symptomatic divided by Asymptomatic

6. Secondary Outcome: Relationship Between End of Day Comfort Scores and Tear Film Osmolarity (Part1: Dailies Aqua Comfort Plus)
Description: Clinical measures (LMS, NIBUT, TMH, tear film osmolarity) were assessed at Visit 4 (14 Hours Follow-up), while density of white blood cells were assessed at Visit 2 (2 week follow-up). Clinical Measures, LMS, NIBUT, TMH and Tear Film Osmolarity were measured in the right (OD) eye only, while white blood cells were assessed in both eyes for both the upper and lower eye lids. End of the day comfort was assessed at Visit 4 for Clinical measures (LMS, NIBUT, TMH, tear film osmolarity), approximately 14 Hours after lens insertion at Visit 3. Visit 3 could occur between two to 180 days after Visit 2. End of Day Comfort for white blood cells was assessed at Visit 2 (2-week after Visit 1). End of the day comfort was assessed using a visual analogue scale (VAS) ranging from 0 - 100, where 0 is uncomfortable and 100 is comfortable. The average end of the day comfort score was reported for the Test 1 (Dailies Aqua Comfort Plus).
Time Frame: VAS, and Tear Film Osmolarity 14 Hours Follow-up at Visit 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Groups:
- Test 1 (Dailies Aqua Comfort Plus): Subjects wore the Test 1 [Dailies Aqua Comfort Plus] lens during period 1 of the study
Arm/Group | Test 1 (Dailies Aqua Comfort Plus)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 76.24 (23.999)
Statistical Analysis 1: Comparison: Test 1 (Dailies Aqua Comfort Plus); Test type: Other — Statistical significance correlation: Statistically Significant correlations were concluded if the upper CL is below 0 or the lower CL is above 0; p = 0.3446, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.1416, 95% CI 2-sided [-0.4148 to 0.1551]

7. Secondary Outcome: Relationship Between End of Day Comfort Scores and Tear Meniscus Height (Part1: Dailies Aqua Comfort Plus)
Description: as for outcome 6
Time Frame: VAS, and TMH 14 Hours Follow-up at Visit 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 1 (Dailies Aqua Comfort Plus)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 76.24 (23.999)
Statistical Analysis 1: Comparison: Test 1 (Dailies Aqua Comfort Plus); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.5556, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = 0.0887, 95% CI 2-sided [-0.2070 to 0.3694]

8. Secondary Outcome: Relationship Between End of Day Comfort Scores and Lid Margin Staining (Part1: Dailies Aqua Comfort Plus)
Description: as for outcome 6
Time Frame: VAS, and Lid Margin staining 14 Hours Follow-up at Visit 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 1 (Dailies Aqua Comfort Plus)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 76.24 (23.999)
Statistical Analysis 1: Comparison: Test 1 (Dailies Aqua Comfort Plus); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.1676, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.2052, 95% CI 2-sided [-0.4676 to 0.0905]

9. Secondary Outcome: Relationship Between End of Day Comfort Scores and Non-invasive Tear Break-up Time (Part1: Dailies Aqua Comfort Plus)
Description: Clinical measures (LMS, NIBUT, TMH, tear film osmolarity) were assessed at Visit 4, (14 Hours Follow-up), while density of white blood cells were assessed at Visit 2 (2 week follow-up). Clinical Measures, LMS, NIBUT, TMH and Tear Film Osmolarity were measured in the right (OD) eye only, while white blood cells were assessed in both eyes for both the upper and lower eye lids. End of the day comfort was assessed at Visit 4 for Clinical measures (LMS, NIBUT, TMH, tear film osmolarity), approximately 14 Hours after lens insertion at Visit 3. Visit 3 could occur between two to 180 days after Visit 2. End of Day Comfort for white blood cells was assessed at Visit 2 (2-week after Visit 1). End of the day comfort was assessed using a visual analogue scale (VAS) ranging from 0 - 100, where 0 is uncomfortable and 100 is comfortable. The average end of the day comfort score was reported for the Test 1 (Dailies Aqua Comfort Plus).
Time Frame: VAS, and NIBUT 14 Hours Follow-up at Visit 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 1 (Dailies Aqua Comfort Plus)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 76.24 (23.999)
Statistical Analysis 1: Comparison: Test 1 (Dailies Aqua Comfort Plus); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.5483, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = 0.0903, 95% CI 2-sided [-0.2054 to 0.3709]

10. Secondary Outcome: Relationship Between End of Day Comfort Scores and Density of White Blood Cells Lower Lid (Part1: Dailies Aqua Comfort Plus)
Description: as for outcome 6
Time Frame: VAS, and WBC before lens removal 6 Hours Follow-up at Visit 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 1 (Dailies Aqua Comfort Plus)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 67.05 (30.322)
Statistical Analysis 1: Comparison: Test 1 (Dailies Aqua Comfort Plus); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.0719, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.2679, 95% CI 2-sided [-0.5205 to 0.0278]

11. Secondary Outcome: Relationship Between End of Day Comfort Scores and Density of White Blood Cells Upper Lid (Part1: Dailies Aqua Comfort Plus)
Description: as for outcome 6
Time Frame: VAS, and WBC before lens removal 6 Hours Follow-up at Visit 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 1 (Dailies Aqua Comfort Plus)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 67.05 (30.322)
Statistical Analysis 1: Comparison: Test 1 (Dailies Aqua Comfort Plus); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.0190, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.3434, 95% CI 2-sided [-0.5786 to 0.0554]

12. Secondary Outcome: Relationship Between End of Day Comfort Scores and Tear Film Osmolarity (Part2: Acuvue Oasys 1-Day)
Description: Clinical measures (LMS, NIBUT, TMH, tear film osmolarity) were assessed at Visit 8 (14 Hours Follow-up), while density of white blood cells were assessed at Visit 6 (2 week follow-up). Clinical Measures, LMS, NIBUT, TMH and Tear Film Osmolarity were measured in the right (OD) eye only, while white blood cells were assessed in both eyes for both the upper and lower eye lids. End of the day comfort was assessed at Visit 8 for Clinical measures (LMS, NIBUT, TMH, tear film osmolarity), approximately 14 Hours after lens insertion at Visit 7. Visit 7 could occur between two to 180 days after Visit 6. End of Day Comfort for white blood cells was assessed at Visit 6 (2-week after Visit 5). End of the day comfort was assessed using a visual analogue scale (VAS) ranging from 0 - 100, where 0 is uncomfortable and 100 is comfortable. The average end of the day comfort score was reported for the Test 2 (Acuvue Oasys 1-Day).
Time Frame: VAS, and Tear Film Osmolarity 14 Hours Follow-up at Visit 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Groups:
- Test 2 (Acuvue Oasys 1-Day): Subjects wore the Test 2 [Acuvue Oasys 1-Day] lens during period 2 of the study
Arm/Group | Test 2 (Acuvue Oasys 1-Day)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 85.28 (18.439)
Statistical Analysis 1: Comparison: Test 2 (Acuvue Oasys 1-Day); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.0420, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.2975, 95% CI 2-sided [-0.5410 to -0.0078]

13. Secondary Outcome: Relationship Between End of Day Comfort Scores and Tear Meniscus Height (Part2: Acuvue Oasys 1-Day)
Description: as for outcome 12
Time Frame: VAS, and TMH 14 Hours Follow-up at Visit 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 2 (Acuvue Oasys 1-Day)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 85.28 (18.439)
Statistical Analysis 1: Comparison: Test 2 (Acuvue Oasys 1-Day); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.3973, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = 0.1270, 95% CI 2-sided [-0.1696 to 0.4024]

14. Secondary Outcome: Relationship Between End of Day Comfort Scores and Lid Margin Staining (Part2: Acuvue Oasys 1-Day)
Description: Clinical measures (LMS, NIBUT, TMH, tear film osmolarity) were assessed at Visit 8 (14 Hours Follow-up), while density of white blood cells were assessed at Visit 6 (2 week follow-up). Clinical Measures, LMS, NIBUT, TMH and Tear Film Osmolarity were measured in the right (OD) eye only, while white blood cells were assessed in both eyes for both the upper and lower eye lids. End of the day comfort was assessed at Visit 8 for Clinical measures (LMS, NIBUT, TMH, tear film osmolarity), approximately 14 Hours after lens insertion at Visit 7. Visit 7 could occur between two to 180 days after Visit 2. End of Day Comfort for white blood cells was assessed at Visit 6 (2-week after Visit 5). End of the day comfort was assessed using a visual analogue scale (VAS) ranging from 0 - 100, where 0 is uncomfortable and 100 is comfortable. The average end of the day comfort score was reported for the Test 2 (Acuvue Oasys 1-Day).
Time Frame: VAS, and LMS 14 Hours Follow-up at Visit 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 2 (Acuvue Oasys 1-Day)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 85.28 (18.439)
Statistical Analysis 1: Comparison: Test 2 (Acuvue Oasys 1-Day); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.8894, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.0210, 95% CI 2-sided [-0.3094 to 0.2710]

15. Secondary Outcome: Relationship Between End of Day Comfort Scores and Non-invasive Tear Break-up Time (Part2: Acuvue Oasys 1-Day)
Description: as for outcome 12
Time Frame: VAS, and LMS 14 Hours Follow-up at Visit 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 2 (Acuvue Oasys 1-Day)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 85.28 (18.439)
Statistical Analysis 1: Comparison: Test 2 (Acuvue Oasys 1-Day); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.6129, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = 0.0762, 95% CI 2-sided [-0.2190 to 0.3585]

16. Secondary Outcome: Relationship Between End of Day Comfort Scores and White Blood Cells Lower Lid (Part2: Acuvue Oasys 1-Day)
Description: as for outcome 12
Time Frame: VAS, and WBC before lens removal at Visit 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 2 (Acuvue Oasys 1-Day)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 85.53 (20.803)
Statistical Analysis 1: Comparison: Test 2 (Acuvue Oasys 1-Day); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.3493, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.1402, 95% CI 2-sided [-0.4137 to 0.1565]

17. Secondary Outcome: Relationship Between End of Day Comfort Scores and White Blood Cells Upper Lid (Part2: Acuvue Oasys 1-Day)
Description: Clinical measures (LMS, NIBUT, TMH, tear film osmolarity) were assessed at Visit 8, (14 Hours Follow-up), while density of white blood cells were assessed at Visit 6 (2 week follow-up). Clinical Measures, LMS, NIBUT, TMH and Tear Film Osmolarity were measured in the right (OD) eye only, while white blood cells were assessed in both eyes for both the upper and lower eye lids. End of the day comfort was assessed at Visit 8 for Clinical measures (LMS, NIBUT, TMH, tear film osmolarity), approximately 14 Hours after lens insertion at Visit 7. Visit 7 could occur between two to 180 days after Visit 6. End of Day Comfort for white blood cells was assessed at Visit 6 (2-week after Visit 5). End of the day comfort was assessed using a visual analogue scale (VAS) ranging from 0 - 100, where 0 is uncomfortable and 100 is comfortable. The average end of the day comfort score was reported for the Test 2 (Acuvue Oasys 1-Day).
Time Frame: VAS, and WBC before lens removal at Visit 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Units Other Than Participants: Eyes
Arm/Group | Test 2 (Acuvue Oasys 1-Day)
Number analyzed (Participants) | 46
Number analyzed (Eyes) | 92
Units on a Scale | 85.53 (20.803)
Statistical Analysis 1: Comparison: Test 2 (Acuvue Oasys 1-Day); Test type: Other — [test comment as in outcome 6, analysis 1]; p = 0.4270, Pearson correlation; Pearson correlation statistics using Fisher's z transformation; Correlation Coefficient = -0.1192, 95% CI 2-sided [-0.3958 to 0.1772]

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The average completion time was 171 days per subject. The minimum completion time was 57 days, and the maximum was 576 days.
Arm/Group | Test 1 (Dailies Aqua Comfort Plus) | Test 2 (Acuvue Oasys 1-Day)
All-Cause Mortality (participants affected / at risk) | 0/184 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/48
Other Adverse Events (participants affected / at risk) | 0/184 | 0/48

LIMITATIONS AND CAVEATS:
Participants were classified as symptomatic or asymptomatic based on their responses to the CLDEQ-8 questionnaire after 2-weeks of lens wear. CLDEQ is a validated questionnaire assessing patient experience of symptoms related to contact lens dryness. Total Scores were calculated by summing subjects' responses to individual items (Chalmers et al, Contact Lens & Anterior Eye 2016, 342-352). Total scores range from 0 to 37 where higher scores indicate more dryness related to contact lens wear.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03871543/Prot_SAP_000.pdf